CLINICAL TRIAL: NCT06400225
Title: MATCH Treatment Subprotocol Z1L: BVD-523FB (Ulixertinib) in Patients With Tumors With BRAF Fusions, or With Non-V600E, Non-V600K BRAF Mutations
Brief Title: Testing BVD-523FB (Ulixertinib) as Potentially Targeted Treatment in Cancers With Genetic Changes (MATCH - Subprotocol Z1L)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2024-01160; NCI-2024-01160 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAY131-Z1L (Other: ECOG-ACRIN Cancer Research Group); EAY131-Z1L (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2024-05-03; First posted 2024-05-06 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Advanced Lymphoma; Advanced Malignant Solid Neoplasm; Refractory Lymphoma; Refractory Malignant Solid Neoplasm; Refractory Multiple Myeloma
MeSH Terms: conditions — Lymphoma; Multiple Myeloma | interventions — Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; Nuclear Medicine Department, Hospital; ulixertinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (BVD-523FB [ulixertinib]) (Experimental): Patients receive BVD-523FB (ulixertinib) PO BID on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo CT or MRI and blood sample collection throughout the trial. Patients also undergo ECHO or nuclear study (MUGA or similar scan) during screening and on study. Patients may also undergo biopsies on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Procedure: Radionuclide Imaging; Drug: Ulixertinib

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Radionuclide Imaging — Undergo nuclear study
  Other Names: NM; Nuclear Medicine; nuclear medicine scan; radioimaging; Radionuclide Scanning; Scan; Scintigraphy
Drug: Ulixertinib — Given PO
  Other Names: BVD-523; VRT752271

SUMMARY:
This phase II MATCH treatment trial tests how well BVD-523FB (ulixertinib) works in treating patients with cancer that has certain genetic changes. BVD-523FB (ulixertinib) is used in patients whose cancer has a mutated (changed) form of a gene called BRAF. It is in a class of medications called kinase inhibitors. It works by blocking the action of proteins that signal cancer cells to multiply. This helps slow or stop the spread of cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the proportion of patients with objective response (OR) to targeted study agent(s) in patients with advanced refractory cancers/lymphomas/multiple myeloma.

SECONDARY OBJECTIVES:

I. To evaluate the proportion of patients alive and progression free at 6 months of treatment with targeted study agent in patients with advanced refractory cancers/lymphomas/multiple myeloma.

II. To evaluate time until death or disease progression. III. To identify potential predictive biomarkers beyond the genomic alteration by which treatment is assigned or resistance mechanisms using additional genomic, ribonucleic acid (RNA), protein and imaging-based assessment platforms.

IV. To assess whether radiomic phenotypes obtained from pre-treatment imaging and changes from pre- through post-therapy imaging can predict objective response and progression free survival and to evaluate the association between pre-treatment radiomic phenotypes and targeted gene mutation patterns of tumor biopsy specimens.

OUTLINE:

Patients receive BVD-523FB (ulixertinib) orally (PO) twice daily (BID) on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo computed tomography (CT) or magnetic resonance imaging (MRI) and blood sample collection throughout the trial. Patients also undergo echocardiography (ECHO) or nuclear study (multigated acquisition [MUGA] or similar scan) during screening and on study. Patients may also undergo biopsies on study.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have met applicable eligibility criteria in the Master MATCH Protocol EAY131/ NCI-2015-00054 prior to registration to treatment subprotocol
* Patients must fulfill all eligibility criteria of MATCH Master Protocol at the time of registration to treatment step (Step 1, 3, 5, 7)
* Patients must have a BRAF non-V600 mutation or BRAF fusion, or another BRAF aberration, as determined via the MATCH Master Protocol
* Patients with BRAF V600E/K/R/D mutations are excluded
* Patients must have an electrocardiogram (ECG) within 8 weeks prior to treatment assignment and must have no clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g. complete left bundle branch block, third degree heart block)
* Patients must not have known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to BVD-523FB (ulixertinib), dimethyl sulfoxide (DMSO), or excipients
* Patients must not have a left ventricular ejection fraction (LVEF) < the institutional lower limit of normal (LLN) or < 50% (whichever is higher)
* Patients must not have prior use of MEK or ERK 1/2 inhibitors
* Patients must not have a history of retinal vein occlusion (RVO) or central serous retinopathy. Patients with visible retinal pathology as assessed by ophthalmologic exam that is considered a risk factor for retinal vein thrombosis or central serous retinopathy will be excluded
* Intraocular pressure is ≤ 21mm Hg as measured by tonography. Patients diagnosed with glaucoma within 1 month prior to Step 1 registration are excluded
* Patients must not have leptomeningeal metastases or spinal cord compression due to disease
* Patients must not have primary malignancy of the central nervous system

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2019-07-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 3 years
  ORR is defined as the percentage of patients whose tumors have a complete or partial response to treatment among analyzable patients. Objective response is defined consistent with Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. 90% two-sided confidence interval is calculated for ORR. For the purposes of this study, patients should be re-evaluated for response:
  * For treatments given in 21 day (3 week) cycles: every 3 cycles (9 weeks) for the first 33 cycles, and every 4 cycles thereafter (12 weeks)
  * For treatments given in 28 day (4 week) cycles: every 2 cycles (8 weeks) for the first 26 cycles, and every three cycles thereafter (12 weeks)
  * For treatments given in 42 day (6 week) cycles: every 2 cycles (12 weeks)

SECONDARY OUTCOMES:
Overall survival (OS) | From start of treatment on that step until death, or censored at the date of last contact, assessed up to 3 years
  Will be evaluated specifically for each drug (or step). OS will be estimated using the Kaplan-Meier method.
6-month progression free survival (PFS) rate | From start of treatment on that step until determination of disease progression or death from any cause, censored at the date of last disease assessment for patients who have not progressed, assessed at 6 months
  Progression free survival is defined as time from treatment start date to date of progression or death from any cause, whichever occurs first. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Please refer to the protocol for detailed definitions of disease progression. 6 month PFS rate was estimated using the Kaplan-Meier method, which can provide a point estimate for any specific time point.
Progression free survival | From start of treatment on that step until determination of disease progression or death from any cause, censored at the date of last disease assessment for patients who have not progressed, assessed up to 3 years
  PFS was defined as time from treatment start date to date of disease progression or death from any causes, whichever occurred first. Median PFS was estimated using the Kaplan-Meier method. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Please refer to the protocol for detailed definitions of disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Subbiah, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (1):
- ECOG-ACRIN Cancer Research Group, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm